CLINICAL TRIAL: NCT04938011
Title: A Randomized Controlled Study of Prolonging the Time of Progesterone Supplementation to Improve the Pregnancy Outcome of Single Day 6 Blastocyst Transfer of Freeze-thaw Cycle
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, Reproductive Medicine Center of The Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SZ-2021-0616
Record Dates: First submitted 2021-06-19; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Progesterone + 7 (Experimental): the transfer of day 6 blastocyst on the 7th day of progesterone supplementation
  Interventions: Drug: progesterone
- Progesterone + 6 (Active Comparator): the transfer of day 6 blastocysts on the 6th day of progesterone supplementation
  Interventions: Drug: progesterone

INTERVENTIONS:
Drug: progesterone — the transfer of day 6 blastocyst on the 6th day of progesterone supplementation
  Arms: Progesterone + 6
Drug: progesterone — the transfer of day 6 blastocyst on the 7th day of progesterone supplementation
  Arms: Progesterone + 7

SUMMARY:
This is a single-center, prospective, randomized controlled study. Patients with single blastocyst transfer in the freeze-thaw cycle, aged from 20 to 38 years, with less than three transfers, and with HRT-cycle single D6 blastocyst transfer in the current cycle were enrolled as the study participants. They were randomized into two groups using an Excel table, and the efficacy was evaluated in a blinded manner by a third party who was unaware of the grouping; the data summary phase was performed by blinded statistical analysis with triple separation of the investigator, operator, and statistician.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20 to 38 years.
2. Less than three transfers.
3. Undergoing HRT freeze-thaw cycle single blastocyst transfer in the current cycle.
4. Having consented to participate in this study and signed the informed consent form.

Exclusion Criteria:

1. Chromosomal abnormality in either the patient or their partner
2. Contraindications to hormone replacement therapy.
3. Patients with intramural myoma affecting the morphology of the uterine cavity, severe adenomyosis, endometriosis, congenital uterine anomalies, endometrial tuberculosis, intrauterine adhesion and other diseases significantly affecting embryonic implantation.
4. Currently participating in another clinical study.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Embryo implantation rate | 30 days after embryo transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Center, The affiliated Drum Towel Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Xu M, Yan Y, Shen X, Sun H, Yan G, Kong N, Jiang Y. Prolonging the time of progesterone supplementation to improve the pregnancy outcomes of single day 6 blastocyst transfer in frozen-thawed cycles: study protocol for a randomized controlled trial. Trials. 2022 Dec 19;23(1):1024. doi: 10.1186/s13063-022-07013-1. PMID 36536470